CLINICAL TRIAL: NCT06042218
Title: New Back. Analysis of the Acute and Chronic Effects of a Program of Body and Postural Work Through "Xiaxi Aligns Your Health"
Brief Title: Xiaxi Program for Back Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Collaborators: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Raquel Vaquero-Cristóbal, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UALBIO2023/005
Record Dates: First submitted 2023-09-04; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Adults; No Sagittal Spine Disposition Disorder; No Surgery on the Spine or the Hamstring; No Specific Treatment for Spinal Pathology; Not Involved in Structured Exercise Programs Before or During the Time of the Study

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group who trained one day a week (Experimental): This intervention group will attend a weekly sixty-minute training session with the Xiaxi machine during the twelve weeks of the intervention. The sessions will include flexibility and strength-resistance work, as well as postural awareness.
  Interventions: Behavioral: Xiaxi intervention program
- Experimental group who trained two days a week (Experimental): This intervention group will attend two weekly sixty-minute training sessions with the Xiaxi machine during the twelve weeks of the intervention. The sessions will include flexibility and strength-resistance work, as well as postural awareness.
  Interventions: Behavioral: Xiaxi intervention program
- Control Group (No Intervention): They will not attend any type of intervention. They will continue to perform their daily activities without intervention.

INTERVENTIONS:
Behavioral: Xiaxi intervention program — The Xiaxi sessions will follow the same structure in both intervention groups. First of all, 8-minute warm-up where the participants will work on: postural awareness; active static stretching of the pectoral, hamstring and psoas muscles; and mobility. The main part will include the following blocks of content during the 12 weeks of intervention (46 minutes will be spent on this part in each session): breathing; mobility; active and dynamic static stretching of the tonic muscles with effects on the spine dynamic; strength of the phasic muscles with effects on the spine dynamic, alternating upper limb, lower limb and core; postural awareness; and passive static stretching of the tonic muscles with effects on the spine dynamic. The cool down will be similar in each session (6 minutes) and will focus on: postural awareness and passive static stretching of the pectoral, hamstring and psoas muscles.
  Arms: Experimental group who trained one day a week; Experimental group who trained two days a week

SUMMARY:
Progressive deformity from the optimal spinal curvatures is a degenerative disorder related to progressive ageing that affects an increasing number of adults. This is one of the main affectations on the health of adults, being its cause multifactorial. That is why a totally effective intervention has not yet been found that allows obtaining a substantial improvement in all the adults who suffer from it. However, certain physical programs that include mind-body work have been effective, but research is limited and the results are inconclusive. For this reason, this research arises, in which a training protocol has been designed using an instrument called Xiaxi with which the body-mind work is prioritized.

The aims of this study were: 1) to evaluate the effects of a 12-weeks Xiaxi® exercise program on the sagittal spinal disposition and hamstring extensibility of adults, and 2) to determine whether the weekly training frequency influenced the changes found on sagittal spinal disposition and hamstring extensibility with Xiaxi® training program.

The present investigation is composed of two data collections that will be carried out before and after a twelve-week intervention. Two intervention groups and a control group make up the sample, with one of the intervention groups attending Xiaxi training once a week and the other intervention group twice a week. The control group will only attend the measurements, but will not participate in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* adults from 20 to 60 years-old
* not have a doctor-diagnosed sagittal spine disposition disorder
* not have had surgery on the spine or the hamstring musculature
* not being under a specific treatment for spinal pathology
* not involve in structured exercise programs before or during the time of the study

Exclusion Criteria:

* not being able to complete all the evaluations
* for members of the experimental group missing more than 20% of the sessions

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-12-08 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Sagittal spinal curvature in relaxed standing | Up to 12 weeks
  The thoracic angle, lumbar angle and pelvic tilt will be measured with the subject in a standing position, adopting the usual and daily position. The unit of measurement will be the same, using the grades achieved.
Sagittal spinal curvature in active alignment in standing | Up to 12 weeks
  The thoracic angle, lumbar angle and pelvic tilt will be measured with the subject in a standing position, but in this case the subject will be asked to rectify the arrangement of the spine to be as straight as possible. The unit of measurement will be the same, using the grades achieved.
Sagittal spinal curvature in relaxed sitting | Up to 12 weeks
  The thoracic angle, lumbar angle and pelvic tilt will be measured with the subject in a seated position, maintaining a habitual, everyday position. The unit of measurement will be the same, using the grades achieved.
Sagittal spinal curvature during Macrae & Wright test | Up to 12 weeks
  The thoracic angle, lumbar angle and pelvic tilt will be measured with the subject performing the Macrae & Wright test, in which the subject will be asked to perform maximum trunk flexion from a seated position. The unit of measurement will be the same, using the grades achieved.
Sagittal spinal curvature during sit and reach test. | Up to 12 weeks
  The thoracic angle, lumbar angle and pelvic tilt will be measured with the subject performing the sit and reach test, in which the subject will be asked to perform a maximum trunk flexion from a seated position and with the soles of the feet resting on a box, keeping the knees fully extended during the same, to push a ribbon the maximum distance through the box. The unit of measurement will be the degrees of the curvatures of the back, as well as the distance reached in the test.
Sagittal spinal curvature during toe touch test | Up to 12 weeks
  The thoracic angle, lumbar angle and pelvic tilt will be measured with the subject performing the toe touch test. In this test, the subject will be asked to perform a maximum trunk flexion in which he/she will try to reach the maximum possible distance from a standing position on a box. The knees will be kept fully extended during the test and an attempt will be made to reach the feet, and this distance may be exceeded if necessary. The unit of measurement will be the degrees of the curvatures of the back, as well as the distance reached in the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No